CLINICAL TRIAL: NCT01098578
Title: Floseal Posterior Epistaxis Pilot Study (PEPIS)
Brief Title: Floseal Treatment for Posterior Epistaxis Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Baxter BS09-000313; REB 2009428-01H (Other: Ottawa Hospital Research Ethics Board)
Record Dates: First submitted 2010-04-01; First posted 2010-04-02 (Estimated); Results first posted 2015-01-26 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Epistaxis
Keywords: Posterior Epistaxis
MeSH Terms: conditions — Epistaxis | interventions — FloSeal Matrix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Floseal (Experimental): Received 1 syringe of Floseal for treatment of posterior epistaxis.
  Interventions: Drug: Floseal

INTERVENTIONS:
Drug: Floseal — Received 1 syringe of Floseal as treatment for posterior epistaxis.
  Other Names: non applicable

SUMMARY:
Effectiveness of Floseal for the treatment of posterior epistaxis.

DETAILED DESCRIPTION:
Floseal, a hemostatic agent, is an effective treatment for anterior epistaxis as well as numerous other acute bleeding conditions throughout the body. The investigators hypothesize that Floseal is an effective treatment for posterior epistaxis. If so, then this will also lead to significant cost savings in comparison to any other method of treatment of posterior epistaxis. The investigators have planned a prospective, nonblinded, nonrandomised study with a total of 40 subjects with posterior epistaxis to be included in this study.

ELIGIBILITY:
Inclusion Criteria:

* age greater than 18 years of age
* posterior epistaxis

Exclusion Criteria:

* patients with anterior epistaxis
* known sensitivity to any of the materials of Floseal or the topical medications administered as part of the evaluation and treatment of epistaxis (lidocaine, xylometazoline hydrochloride)
* pregnant or breast feeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-04; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shaun Kilty, MD, Principal Investigator — Ottawa Hospital Research Institute

REFERENCES:
- [Derived] Kilty SJ, Al-Hajry M, Al-Mutairi D, Bonaparte JP, Duval M, Hwang E, Tse D. Prospective clinical trial of gelatin-thrombin matrix as first line treatment of posterior epistaxis. Laryngoscope. 2014 Jan;124(1):38-42. doi: 10.1002/lary.24240. Epub 2013 Jun 28. PMID 23754469
- See also: Ottawa Hospital Research Institute — http://www.ohri.ca

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients who presented to the emergency department with posterior epistaxis or who were already admitted to hospital for another diagnosis and had posterior epistaxis were offered enrollment. Recruitment period April 2010- April 2012
Groups:
- Floseal.: Floseal® was used for posterior epistaxis treatment with simultaneous ipsilateral choanal occlusion.
Period: Overall Study
Arm/Group | Floseal.
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Floseal: Received Floseal treatment for posterior epistaxis.
  Floseal : Received Floseal as treatment for posterior epistaxis.
Arm/Group | Floseal
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.8 (20.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 10
Region of Enrollment [Number; unit: participants]
  Canada | 20

OUTCOME MEASURES:

1. Primary Outcome: Effectiveness of Floseal for the Treatment of Posterior Epistaxis.
Description: Successful treatment using the gelatin-thrombin matrix protocol (Floseal) was any case of posterior epistaxis that stopped following the immediate application of either one or two syringes of Floseal® and the epistaxis did not resume within fourteen days of the treatment date.
Time Frame: Immediate effect with 1 hour observation and follow-up at 5 and 30 days following treatment.
Measure: Number; unit: participants
Arm/Group | Floseal
Number analyzed (Participants) | 20
participants | 20

2. Secondary Outcome: Cost Savings of Floseal Treatment in Comparison to Posterior Packing, Surgical, and Embolisation Treatments for Posterior Epistaxis.
Description: The institutional cost for the treatment of posterior epistaxis patients with posterior packing, endoscopic surgery, and endovascular embolization, at TOH were calculated and compared with the institutional cost of a patient visit for posterior epistaxis successfully treated with the study protocol using Floseal. All costs were calculated in Canadian dollars (CAD), they were converted to US dollars (USD) using the current monetary exchange rate (total CAD x 1.03= total USD). For all of the patients treated in this study, the total institution cost was $24487.53 (USD). The minimal institutional cost of successfully treating all of the study patients with endoscopic surgery, would have been $53933.89 (USD) or 2.2 times the actual expense. (Total cost 20 participants Floseal/expected total cost 20 endoscopic surgery*100)This represents savings of $29446.39 (USD) or 45.40%
Time Frame: 30 days
Measure: Number; unit: percentage of expected cost
Arm/Group | Floseal
Number analyzed (Participants) | 20
percentage of expected cost | 45.40

3. Other Pre Specified Outcome: Total Institutional Cost Savings
Description: Difference between the total institutional cost of successfully treating 20 study patients with Floseal compared to the total institutional cost of treating the same number of patient with endoscopic surgery
Time Frame: End of study. Cost calculated after 20 patients were treated with Floseal
Measure: Number; unit: US Dollars
Groups:
- FLOSEAL: Institutional cost of treating all study patients with Floseal for posterior epistaxis
- Endoscopic Surgery: The calculated minimal institutional cost if all the study patients had been treated with endoscopic surgery for posterior epistaxis
Arm/Group | FLOSEAL | Endoscopic Surgery
Number analyzed (Participants) | 20 | 20
US Dollars | 24487.53 | 53933.89

ADVERSE EVENTS:
Time Frame: Adverse events were evaluated from the time of treatment with Floseal and up to 30 30 days after treatment with Floseal
Arm/Group | Floseal
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes